CLINICAL TRIAL: NCT03161392
Title: Evaluation of Solitary Dilated Duct Visualized by Mammography in Correlation With Ultrasonography and Anatomopathological Findings.
Brief Title: Correlation of Solitary Dilated Duct at Mammography With Ultrasonography and Anatomopathological Findings
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina do ABC (Other)
Collaborators: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Luciano de Melo Pompei', Professor, Faculdade de Medicina do ABC
Other Study IDs: Ductoisolado_01
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Mammary Duct Ectasia of Unspecified Breast; Mammographic Findings; Female
Keywords: mammography; ductal ectasia; breast neoplasm/diagnostic imaging; mammary Glands, Human/pathology; female
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ductal lesion: Subjects with a ductal lesion detected on ultrasonography.
  Interventions: Diagnostic Test: Ultrasound-guided percutaneous biopsy
- No ductal lesion: Subjects without a ductal lesion detected on ultrasonography
  Interventions: Diagnostic Test: Follow-up

INTERVENTIONS:
Diagnostic Test: Follow-up — Group "No ductal lesion" will be submitted to follow-up with periodic breast ultrasonography/mammography every 6 months for 2 years.
  Groups: No ductal lesion
Diagnostic Test: Ultrasound-guided percutaneous biopsy — Group "Ductal lesion" will be submitted to ultrasound-guided percutaneous biopsy and the specimen will be histologically analysed.
  Groups: Ductal lesion

SUMMARY:
Mammograms performed at the Diagnostic Imaging Department of the "Instituto Brasileiro de Controle do Câncer" (IBCC - Brazilian Cancer Control Institute) will be prospectively evaluated. Patients who present a solitary dilated duct visualized by mammography will be submitted to breast ultrasonography. In case of detection of lesion, a percutaneous biopsy will be performed.

DETAILED DESCRIPTION:
Purpose: To determinate the incidence, pathological significance and risk factors associated with the presence of solitary dilated duct visualized at mammography exam.

Methods: Mammograms performed at the Diagnostic Imaging Department of the "Instituto Brasileiro de Controle do Câncer" (IBCC - Brazilian Cancer Control Institute) will be prospectively evaluated. Patients who present a solitary dilated duct visualized by mammography will be included in the study. These patients will be recalled in order to be submitted to an ultrasonography directed to the mammographic finding. Patients who present lesions on ultrasonography will undergo method-guided percutaneous biopsy.

Patients with ductal ectasia, without evident lesions, will be followed for 2 years to evaluate stability by means of mammography or ultrasonography every 6-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Identification of a solitary dilated breast duct at mammography

Exclusion Criteria:

* Previous breast surgery at same side of detection of dilated duct

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women submitted to mammography for breast cancer screening or for diagnosis purposes
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Abnormal histological finding at breast biopsy | At guided-percutaneous biopsy
  Detection of any histological abnormality

CONTACTS AND LOCATIONS:
Overall Officials: Luciano M Pompei, PhD, Study Director — ABC Medicine School

IPD SHARING:
Plan to Share IPD: No